CLINICAL TRIAL: NCT03245164
Title: Comparing the Effects of Group Exercise and Basketball on Body Composition and Motor Skills of Obese Children
Brief Title: The Effects of Group Exercise and Basketball on Obese Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Mediterranean University (Other)
Collaborators: Hacettepe University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EasternMUZ
Record Dates: First submitted 2017-07-31; First posted 2017-08-10 (Actual); Last update posted 2017-08-10 (Actual); Status verified 2017-08

CONDITIONS: Childhood Obesity; Physical Activity
Keywords: obese children; motor skills; physiotherapy; basketball
MeSH Terms: conditions — Pediatric Obesity; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Physiotherapy group exercises (Experimental): This group continued physiotherapy group exercises for 12 weeks.
  Interventions: Other: Physiotherapy group exercises
- Basketball program (Experimental): Basketball educaiton was presented for 12 weeks.
  Interventions: Other: Basketball program
- Control group (No Intervention): This group did not continue any physical activity regularly.

INTERVENTIONS:
Other: Physiotherapy group exercises — Physiotherapy exercises had aerobic, balance, strength exercises with music.
  Arms: Physiotherapy group exercises
Other: Basketball program — Basketball education presented the techniques about playing basketball and basketball games were played.
  Arms: Basketball program

SUMMARY:
This study aimed to compare the effects of group exercises under physiotherapist control and basketball program on body composition and motor skills of obese children. 45 obese children aged 10 years were randomly included to the physiotherapy (n=15), basketball (n:15), and control group (n:15). The children were assessed before and after 12-week study duration. Body Mass Index (BMI), the percentage of body fat, and circumference values of the children were recorded. Bruininks-Oseretsky Test of Motor Proficiency-Brief Form (BOTMP-BF) was used to determine motor skills of children.

DETAILED DESCRIPTION:
The roles of active physiotherapy programs and sport programs on the management of the problems arising from childhood obesity should be determined. Although the effects of exercise and various sport branches on decrease obesity and obesity related problems, the effects of group exercises managed by physiotherapists and team sports on body composition and motor skills of obese children are not clear so health professionals may have difficulties while suggesting better physical activity for this population.

Thus, body composition and motor skills of the included children were recorded at the beginning. They were then grouped into three in order to compare the effects of group exercises and basketball. Children in the control group did not participate in any of them. Intervention lasted 12 weeks so they were then taken to the assessments at the end of this duration.

ELIGIBILITY:
Inclusion Criteria:

* children who were born in 2006 (10 years old),
* children whose BMI values were ≥95. Percentiles,
* a report which was given by a doctor to state that the child could participate in aerobic exercise,
* children who had not continued to a diet program for 3 months,
* children who had not participated regularly in any sport or exercise for 6 months.

Exclusion Criteria:

* children who had any disease requiring use of medicine,
* children who had any pain to prevent doing exercise or sport,
* children who had any neuromuscular disease

Ages: 10 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Bruininks-Oseretsky Test of Motor Proficiency-Brief Form (BOTMP-BF) | 12 weeks
  The BOTMP-BF test was used to determine the motor skills of the children. It is a popularly used test to specify the level of motor skills of children. Touching nose with index fingers as eyes closed and pivoting thumbs and index fingers were scored for bilateral coordination. Walking forward heel-to-toe on a line for balance, push-up numbers for strength,and number of one-legged side hop in a given duration for speed-agility were scored. Filling in a star, drawing a line through a path, and copying shapes were scored to determine fine motor integration. Stringing blocks in a given time duration was scored for manual dexterity. Catching a Tossed-ball with one hand and dribbling a ball with alternative hands were scored for upper limb coordination. Scoring is explained in the booklet of BOTMP-BF. A total score of this test was acquired.

SECONDARY OUTCOMES:
Body Mass Index | 12 weeks
  Body Mass Index (BMI) was calculated as weight (in kilograms) divided by height (in meters) squared (kg/m2).
Body Fat | 12 weeks
  Body fat was determined by skinfold measurements (in milimeters). Lange Skinfold caliper (Cambridge Scientific Industries, Cambridge, MD) was used to determine the percentage of body fat. Triceps, biceps, chest, sucscapula, abdominal, and suprailiac regions were measured. All measurements were taken only from the right side of their body. During these measurements, all children remained standing. Slaughter's equation was used to calculate the percentage of body fat.
Circumferences | 12 weeks
  Arm, waist, chest, and hip circumferences were measured using an inelastic tape while the children were standing and breathing normally. Right arm was taken as a reference for circumference. Values were recorded in centimeters.

CONTACTS AND LOCATIONS:
Overall Officials: OZLEM ÜLGER, Assist.Prof., Study Director — Hacettepe University

IPD SHARING:
Plan to Share IPD: Yes
Body Mass Indexes of children who continued 4th class in all primary schools in the study city were recorded. The parents of children who had 95.> percentiles of BMI values were then invited to the study and the participants who accepted the invitation were assessed. They were then evaluated and randomly assigned to three groups. The number for each group was determined by power analysis.
Supporting Information: Study Protocol, ICF, CSR, Analytic Code
Time Frame: 2 months
Access Criteria: Primary schools of the city where the study would take place in were analysed for the appropriate body mass indexes. The parents were then invited to participate in the study.

REFERENCES:
- [Background] Alberga AS, Prud'homme D, Sigal RJ, Goldfield GS, Hadjiyannakis S, Phillips P, Malcolm J, Ma J, Doucette S, Gougeon R, Wells GA, Kenny GP. Effects of aerobic training, resistance training, or both on cardiorespiratory and musculoskeletal fitness in adolescents with obesity: the HEARTY trial. Appl Physiol Nutr Metab. 2016 Mar;41(3):255-65. doi: 10.1139/apnm-2015-0413. Epub 2015 Nov 9. PMID 26881317